CLINICAL TRIAL: NCT04298788
Title: Food Intake and Blue Dishware in Residents Living With Dementia in Retirement Homes
Brief Title: Food Intake and Blue Dishware in Residents Living With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Principal Investigator, Heather Keller, Professor, University of Waterloo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ORE40986
Record Dates: First submitted 2020-02-22; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Food Preferences; Eating Behavior
MeSH Terms: conditions — Food Preferences; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: participant meals were randomized to blue or white dishware conditions, matched for food choices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White dishware (Placebo Comparator): standard white dishware used in the home
  Interventions: Other: Blue dishware
- blue dishware (Experimental): specially designed blue dishware, plates and bowls
  Interventions: Other: Blue dishware

INTERVENTIONS:
Other: Blue dishware — blue dishware is used for plates and bowls

SUMMARY:
Blue dishware was alternated with white dishware for lunch and dinner for residents living with dementia. Food consumption occurred in the home dining room and food was weighed before and after consumption to determine proportion consumed. Eating challenges were also noted. Within-participant comparisons were made to determine if food intake and eating challenges improved with the blue dishware condition.

ELIGIBILITY:
Inclusion Criteria:

* living in a residential care environment with dementia
* informed consent of POA and assent of person living with dementia

Exclusion Criteria:

* did not come to the dining room to eat
* required eating assistance
* did not live on the study unit

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Precent of Food consumed of food served (grams consumed/grams provided) | 8 weeks
  gram weight of food intake as weighed on a calibrated scale

SECONDARY OUTCOMES:
Percent of Meals with an Eating challenge based on an Eating challenges Checklist | 8 weeks
  change in eating challenges from a prespecified list

CONTACTS AND LOCATIONS:
Overall Officials: Heather Keller, Principal Investigator — University of Waterloo
Locations (1):
- Riverside Glen, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donnelly R, Wei C, Morrison-Koechl J, Keller H. The effect of blue dishware versus white dishware on food intake and eating challenges among residents living with dementia: a crossover trial. BMC Res Notes. 2020 Jul 23;13(1):353. doi: 10.1186/s13104-020-05195-y. PMID 32703270